CLINICAL TRIAL: NCT01027325
Title: Effects of Resistant Starch on Lipid and Glucose Metabolism in Insulin Resistance
Brief Title: Resistant Starch Insulin Sensitivity Trial
Acronym: RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1RC1DK086472-01 (NIH); 1RC1DK086472-01 (NIH)
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Healthy; Cardiovascular Disease; Atherogenic Dyslipidemia; Insulin Resistance
Keywords: Resistant Starch; Amylose; Amylopectin; LDL subclasses; Dietary carbohydrate; Postprandial insulinemia
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance | interventions — Diet Therapy; Dietary Carbohydrates; Resistant Starch; Amylose; Amylopectin; Lipids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- High CHO/Low Amylose (Experimental): 55% Carbohydrate (11.2% Amylose, 26.3% Amylopectin) 20% Protein 25% Fat
  Interventions: Other: Dietary Intervention
- Low Carbohydrate/Hi Amylose (Experimental): 40% Carbohydrate (26.3% Amylose, 11.2% Amylopectin) 20% Protein 40% Fat
  Interventions: Other: Dietary Intervention
- High CHO/High Amylose (Experimental): 55% Carbohydrate (26.3% Amylose, 11.2% Amylopectin) 20% Protein 25% Fat
  Interventions: Other: Dietary Intervention
- Low Carbohydrate/Low Amylose (Experimental): 40% Carbohydrate (11.2% Amylose, 26.3% Amylopectin) 20% Protein 40% Fat
  Interventions: Other: Dietary Intervention
- Baseline (Active Comparator): 40% Carbohydrate 20% Protein 40% Fat
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Starch digestibility and carbohydrate quantity
  Other Names: Dietary carbohydrate; Resistant starch; Amylose; Amylopectin; Lipids

SUMMARY:
The alarming increase in the prevalence of obesity is a cause of great concern given its association with many adverse health conditions, including insulin resistance and type 2 diabetes, which are associated with increased cardiovascular disease (CVD) risk. The primary objective of this project is to identify effective dietary strategies, focused on carbohydrate quantity and starch digestibility, to improve outcome variables associated with CVD risk in insulin resistant individuals who express components of the atherogenic lipoprotein phenotype (ALP). Current dietary guidelines emphasize substitution of carbohydrate calories for total and saturated fat calories for prevention and management of chronic disease. Yet, we and others have shown that high-carbohydrate diets increase the expression of the ALP, characterized by increased plasma triglycerides, reduced HDL cholesterol, and increased levels of small, dense LDL particles, and that this phenotype is reversed by moderate carbohydrate restriction. We have also shown that expression of stearoyl coenzymeA desaturase (SCD), an enzyme involved in triglyceride synthesis, is reduced with carbohydrate restriction and that this change is correlated with plasma triglyceride response. While carbohydrate restriction is effective for management of ALP, the role of starch quality has not been addressed. Furthermore, there has been no study of the effects of resistant vs. digestible starches incorporated into high- vs. lower carbohydrate diets. Since isolated reports suggest that increased intake of resistant starch lowers plasma triglycerides and postprandial insulinemia, we hypothesize that starch quality is an important determinant of components of ALP, and that this may be mediated in part by reduced adipose tissue SCD expression. Aim 1 and of this proposal will address this hypothesis by a controlled dietary intervention in 52 insulin resistant men and women in which changes in plasma lipids, lipoproteins and lipogenic gene expression will be determined after substituting resistant starch for digestible starch in a high- vs. lower-carbohydrate diet. In Aim 2, the fasting and postprandial glucose and insulin responses to a resistant vs. digestible starch meal will be measured to test the hypothesis that starch digestibility improves glycemic and insulinemic control in a way that relates to diet-induced changes in plasma lipids and lipoproteins.

DETAILED DESCRIPTION:
Clinic Visits:

Participants will visit the clinic a total of 11 times from screen to completion of the study. This will include weekly visits with a dietician and 7 visits requiring blood draws (screen and twice following each diet period). At each visit, participants will be weighed, waist and hip circumferences will be measured, and blood pressure will be monitored. The total amount of blood collected is 450ml.

Screening visit (V1: 1 hour):

Recruiters will initially determine eligibility through review of a screening questionnaire and a telephone or personal interview. If a potential subject is eligible and interested, an orientation package will be mailed that will include written information about the study requirements. Interested subjects will be scheduled for a screening visit to determine final eligibility by the Clinical staff. At the screening visit (V1), informed consent will be obtained, anthropometric measurements obtained (height, weight, waist circumference, blood pressure), and blood (30ml) will be drawn to assess laboratory criteria for enrollment (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, glucose, and insulin for determination of HOMA-IR). Screening blood samples from individuals who are either not eligible or unwilling to proceed with the intervention will be destroyed. We will screen for pregnancy, and repeat pregnancy tests after all "A" visits (V2a, v3a, v4a). Menstruating women will be given a calendar to record their menstrual cycle for the duration of the study. Eligible individuals will be contacted within 2 weeks of this screen visit and invited to participate in the study. We are prepared to enroll up to 64 participants in this study to yield a target of 52 completed participants (20% dropout).

Dietitian Visits (Initial: 1 hr, Subsequent: 15 min):

Participants will meet weekly with a dietitian or dietitian aide to receive counseling including weight management and diet review. At these meetings, participants will receive a week's worth of frozen entrees, standardized menus with check lists, and itemized grocery lists. Baked goods and products containing the test starches will also be provided at this time. The form in which they will be provided (frozen or fresh) will depend on the nature of the product and its capacity to withstand refrigerated vs. frozen storage. During the washout period (days 28-42), subjects will continue to refrain from alcohol but will consume their usual home diet for 7 days, followed by the baseline diet for an additional 7 days. We anticipate that giving participants permission to eat what they want for 7 days during the washout will improve their compliance during the remainder of the dietary protocol.

Participants will bring grocery store receipts from the previous week so that the dietitians may ensure purchase of prescribed foods not provided by the Bionutrition Unit.

Post-diet Visits Requiring Blood Draws (A visits: 2.5 hr, B visits: 5 hr):

Participants will visit the clinic on two separate days following completion of each diet to provide blood samples. Duplicate sampling reduces biological variability, and hence improves the power of the study to detect significant diet-induced changes in measurement. On the penultimate day of each diet (Visits 2A, 3A, 4A) participants will visit the clinic in the fasting state and provide a fasting blood sample (30ml) for measurement of total, LDL- and HDL-cholesterol, triglycerides, apolipoproteins A1 and B, and lipoprotein subfraction analysis by ion mobility. Lipoprotein lipase and hepatic lipase activities will also be measured in plasma (20ml) obtained 15 minutes after IV heparin (75 units/kg). On the final day of each diet (Visits 2B, 3B, 4B), participants will provide a second fasting blood sample (for lipids and lipoproteins as above) and an adipose tissue aspiration to measure lipogenic gene expression. In addition a 3 hour starch tolerance meal will be performed at visits 3B and 4B, with blood samples for measuring glucose and insulin drawn in the fasting state and 30, 60, 120, and 180 minutes after a starch meal (60ml total).

Clinical Procedures:

Clinical measurements: Blood pressure will be measured 3 times in a sitting position and the last 2 values averaged. Anthropometric measurements include height, weight, waist and hip circumference, and % body fat by bioimpedance (Tanita scale). Waist circumference is measured two times at the iliac crest and hip circumference is measured at the widest point of the hips.

Standard Blood sampling: Using standard blood collection procedures, blood samples will be collected from participants after a 12-14 hour fast. The blood will be collected into tubes containing the following preservative solution: 3.0 gms EDTA (dipotassium), 1.7 mg P-Pack, 0.15 gms gentamycin sulfate, 0.15 gms chloramphenicol, 5.96 mls aprotinin (Sigma A-6279), and 0.30 gms sodium azide all of which are diluted to 20mls with doubly deionized water. Plasma is separated by immediate centrifugation at 4°C. Lipid and lipoprotein measurements are performed and aliquots of plasma are frozen for future analyses.

Post-heparin Blood Sampling:

A blood sample (20ml) will be drawn 15 minutes after intravenous administration of a heparin bolus (75U/kg, see Risk section for justification) for the analysis of plasma lipase activity. Prior to administration, participants will be interviewed for family history of clotting disorders or personal contraindications including use of anticoagulants, history of bleeding or bruising abnormalities or other diseases, allergies, or recent dental work. Following administration, participants will remain in clinic for 2 hours under observation. They will also be provided with an information sheet regarding heparin and the procedure.

Adipose Tissue Biopsy:

Adipose biopsies will be collected from the subcutaneous flanking region by an R.N. using a standardized, sterile procedure. Participants will be instructed not to take any drugs within 2 days of the procedure that would impair clotting. This procedure will take place at least 24 hours after post-heparin lipase analysis. Because the half-life of heparin is 2 hours, this is sufficient time to ensure clearance. After cleaning the area above the participant's buttock with betadine, Lidocaine hydrochloride 1% (10mg/ml) will be injected into the subcutaneous skin. Using a number 14G needle, 1-1.5 c.c.'s of fat will be aspirated. Cold pressure will be held on site and then the wound will be bandaged. Participants will be instructed to change the bandage once daily for two days. They will be provided with two bandages, instructions for keeping the wound clean, and a telephone number where clinical staff can be reached.

Starch Meal Test:

Immediately following adipose tissue biopsy and fasting blood draw, participants will be given a starch meal that provides 1/3 of the daily calories to be consumed in 15 minutes. It will be similar in macronutrient composition to the test diet to which the participant is assigned and will either be high in amylose or amylopectin. Blood will be drawn 30, 60, 120, and 180 minutes after meal consumption through an IV. For this procedure, an intravenous cannula or needle will be placed in the antecubital vein. A normal saline solution will be run at a keep open rate at the antecubital site.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 20 years
* Blood pressure less than 150/90. If on three separate clinic visits blood pressure remains above this level, a subject will be referred to his or her physician for treatment.
* Body mass index (BMI) ≥ 20 and ≤ 35 kg/m2.
* Non-smoking and does not use nicotine products or recreational drugs.
* Agrees to consume no alcohol or dietary supplements during the study.
* Total cholesterol and LDL cholesterol <95th percentile for sex and age.
* Fasting triglycerides <500mg/dl.
* HOMA-IR ≥ 50th percentile for sex.
* Fasting blood sugar (FBS) < 126 mg/dl.
* Hematocrit ≥ 36%.
* At least 3 months of a weight stable state. During the study, subjects will be required to maintain their body weight within ± 3% (up to a maximum change of 5 lbs) of their initial weight over the course of any consecutive two weeks.
* For women of childbearing potential, two barrier methods of contraception must be used throughout the study and urine pregnancy B-hCG will be done at screen (v1) and at all "A" visits (v2a, 3a, 4a). Subjects who become pregnant will no longer be allowed to continue the study.
* Women will be considered post-menopausal if ≥ 3 years since last menses or no menses for 1-3 years and plasma FSH elevated into postmenopausal range.
* Subjects who cannot complete the requirements of the study for reasons determined by the investigator (i.e. non-accessible veins for blood drawing, inability to keep clinic appointments) will not be able to participate in the study.

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin cancer) in the last 5 years.
* Taking drugs known to affect lipid metabolism, blood thinning agents or hormones
* Abnormal thyroid stimulating hormone (TSH) levels

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 2 weeks, 4 weeks, 8 weeks
LDL subfractions | 2 weeks, 4 weeks, 8 weeks

SECONDARY OUTCOMES:
Total cholesterol | 2 weeks, 4 weeks, 8 weeks
HDL-cholesterol | 2, 4, 8 weeks
apolipoproteins B, AI | 2, 4, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Nathalie Bergeron, PhD, Principal Investigator — Children's Hospital Oakland Research Institiute
Locations (2):
- United States (2):
  - Cholesterol Research Center, Berkeley, California
  - Children's Hospital Oakland Research Institute, Oakland, California